CLINICAL TRIAL: NCT01557296
Title: Comparing Treatment With Food of Small Particle Size and Food of Large Particle Size in Subjects With Diabetic Gastroparesis. Evaluation of Diagnostic Methods. Determination of the Motility of Gastric Emptying After Intervention
Brief Title: Evaluation of Diagnostic Methods and Dietary Treatment of Diabetic Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #EMS-5115#
Record Dates: First submitted 2012-03-16; First posted 2012-03-19 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Diabetic Gastroparesis
Keywords: Diet; Dietary treatment; Particle size; Gastroparesis; Diabetes Mellitus
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — Quality of Life; Nutritional Status; Cell Movement; Gastric Emptying

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetic diet (Placebo Comparator): Control group. Subjects with Insulin Treated Diabetes Mellitus and Gastroparesis. Diet: Food of large particle size during 20 weeks.
  Interventions: Dietary Supplement: dietary treatment: food of small particle size; Radiation: Validate X-ray diagnostic method.; Other: Can the motility be improved; Biological: postprandial plasma glucose
- Diet food in small particle size (Active Comparator): Intervention group: Subjects with Insulin Treated Diabetes and Gastroparesis. Intervention Diet: Food of small particle size during 20 weeks.
  Interventions: Dietary Supplement: dietary treatment: food of small particle size; Radiation: Validate X-ray diagnostic method.; Other: Can the motility be improved; Biological: postprandial plasma glucose

INTERVENTIONS:
Dietary Supplement: dietary treatment: food of small particle size — Subjects with diabetes mellitus and gastroparesis. Insulin treatment. Dietary treatment with food of small particle size.
  Other Names: Randomized study; Diabetic gastroparesis; Dietary treatment:Food of small particle size; Metabolic control; Gastrointestinal symptoms; Quality of life; Nutrition status; Autonomic neuropathy
Radiation: Validate X-ray diagnostic method. — Follow 20 radiopaque markers throw the ventricle by X-ray.
  Other Names: Radiopaque markers method; Gastric scintigraphy
Other: Can the motility be improved — Registered the gastric emptying after intervention. Comparing the registrations at the beginning and at the end of the study.
  Other Names: motility; gastric emptying; improved gastric emptying
Biological: postprandial plasma glucose — Measure the blood glucose response and gastrointestinal symptoms after a test meal
  Other Names: gastric emptying; plasma glucose response; metabolic control

SUMMARY:
The objective of the study is in subjects with Insulin Treated Diabetes Mellitus type 1 or 2 and gastroparesis:

* validate radiopaque markers with fluoroscopy with gastric scintigraphy method
* study the difference of metabolic control including the frequents of hypoglycaemia, gastrointestinal symptoms, quality of life and nutrition state during dietary treatment of food of small particle size compared with food of large particle size
* validate the radiopaque markers method and measurement of the blood glucose and gastrointestinal symptoms after a test meal, against the gastric scintigraphy
* determine if the function of gastric emptying can be improved after intervention

ELIGIBILITY:
Inclusion Criteria:

* diabetes type 1 or 2 and gastroparesis
* must be able to understand oral and verbal instructions

Exclusion Criteria:

* gastrointestinal surgery
* other gastrointestinal disease
* S-Creatinine >150 umol/L
* mental disease
* cerebral disease
* collagen disease
* untreated endocrine disease
* anticholinergic drugs
* psychopharmacologic drugs
* opiates
* addiction to drugs as alcohol and narcotics
* vegetarian

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Metabolic Control - HbA1c | 22 weeks

SECONDARY OUTCOMES:
gastrointestinal symptoms - Questionnaire: Patient Assessment of upper Gastrointestinal Disorders Symptoms, Gastrointestinal Symptom Rating Scale | 22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Simrén, M.D., Ph.D., Study Chair — Inst of Medicine, Sahlgrenska Academy, Göteborg University
Locations (1):
- Goteborg Universitet, Sahlgrenska Academy, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Olausson EA, Storsrud S, Grundin H, Isaksson M, Attvall S, Simren M. A small particle size diet reduces upper gastrointestinal symptoms in patients with diabetic gastroparesis: a randomized controlled trial. Am J Gastroenterol. 2014 Mar;109(3):375-85. doi: 10.1038/ajg.2013.453. Epub 2014 Jan 14. PMID 24419482